CLINICAL TRIAL: NCT01082146
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [Issthiazolyl-3-14C]-Lurasidone Following Postprandial Single Oral Dose Administration in Health Male Subjects
Brief Title: RI-AME Study OF [ISOTHIAZOLYL-3-14C]-LURASIDONE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1050262
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics; Metabolism
Keywords: pharmacokinetics, lurasidone
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lurasidone (Experimental): LURASIDONE 40mg
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — 40 mg suspension, PO, for 7 days

SUMMARY:
This will be an open-label, non-randomized, absorption, metabolism, and excretion study of Lurasidone administered in a suspension at 40 mg to 6 normal healthy male subjects in a postprandial state

DETAILED DESCRIPTION:
A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [Isothiazolyl-3-14C]-Lurasidone Following Postprandial Single Oral Dose Administration in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. within a BMI range of 18.0 to 28.0 kg/m2 inclusive;
2. males will either be sterile or agree to use from Check-in until 45 days following Study Completion/Discharge approved methods of contraception
3. able to comprehend and willing to sign an Informed Consent Form (ICF);
4. able to void urine on a daily basis and 1 to 2 bowel movements per day.
5. able to swallow 60 mL of dosing suspension.

Exclusion Criteria:

1. history or presence of an abnormal ECG
2. participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in.
3. exposure to significant radiation within 12 months prior to Check-in;
4. participation in any other investigational study drug trial
5. use of any prescription medications/products within 14 days prior to Check-in
6. use of any inhibitors or inducers of CYP3A4 taken within 30 days prior to Check-in, including but not limited to drugs listed in Appendix E;
7. receipt of blood products within 2 months prior to Check-in;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics (PK) of a postprandial single dose of 40 mg (150 Ci 5.55 Megabecquerels (MBq)) [Isothiazolyl-3-14C-Lurasidone and its metabolites | 28 days
To determine the whole blood and serum concentrations of total radioactivity of [Isothiazolyl-3-14C]-Lurasidone (150 Ci). | 28 days
To determine the urinary and fecal recovery of total radioactivity of [Isothiazolyl-3-14C]-Lurasidone (150 Ci). | 28 days

SECONDARY OUTCOMES:
To assess the safety of 40 mg [Isothiazolyl-3-14C]-Lurasidone | 28 days
To characterize and identify metabolites of Lurasidone in serum and urine | 28 days
To determine serum concentrations of Lurasidone | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Bohn, MD, Principal Investigator — Covance Global Clinical Research Unit Inc.
Locations (1):
- Covance Global Clinical Research Unit Inc., Madison, Wisconsin, United States